CLINICAL TRIAL: NCT05459220
Title: A Phase Ⅲ, Randomized, Double-blind, Placebo-controlled Study of SHR0410 Injection for the Treatment of Pain After Laparoscopic Surgery
Brief Title: A Trial of SHR0410 Injection for the Treatment of Pain After Laparoscopic Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR0410-302
Record Dates: First submitted 2022-06-30; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-06

CONDITIONS: Postoperative Pain Of Laparoscopic Surgery

STUDY DESIGN:
Intervention Model Description: SHR0410 injection compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental): SHR0410 Injection（Low Dose）
  Interventions: Drug: SHR0410 Injection
- Treatment group B (Experimental): SHR0410 Injection（High Dose）
  Interventions: Drug: SHR0410 Injection
- Treatment group C (Placebo Comparator): Placebo for SHR0410 Injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR0410 Injection — SHR0410 Injection（Low Dose）
  Arms: Treatment group A
Drug: SHR0410 Injection — SHR0410 Injection（High Dose）
  Arms: Treatment group B
Drug: Placebo — Placebo for SHR0410 Injection.
  Arms: Treatment group C

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of SHR0410 injection for the treatment of pain after laparoscopic surgery

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Subjects requiring elective general anesthesia endoscopic surgery of the lower abdominal
3. Male or female
4. Meet the body mass index standard
5. Conform to the ASA Physical Status Classification

Exclusion Criteria:

1. Subjects with a history of difficult airway
2. Subjects with a history of mental illness
3. Subjects with a history of cognitive impairment epilepsy
4. Subjects with a history of myocardial infarction or unstable angina pectoris
5. Subjects with atrioventricular block or cardiac insufficiency
6. Subjects with a history of ischemic stroke or transient ischemic attack
7. Subjects with poor blood pressure control after medication
8. Subject with a history of substance abuse and drug abuse
9. Abnormal values in liver function
10. Allergic to drugs that may be used during the study
11. Pregnant or nursing women
12. No birth control during the specified period of time
13. Participated in clinical trials of other drugs (received experimental drugs)
14. The investigators determined that other conditions were inappropriate for participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Summed Pain Intensity Difference From 0-24 Hours (SPID0-24) | 0 to 24 hours
  Pain intensity will be evaluated using an 11-point (0-10) numeric rating scale (NRS), with higher numbers indicating a higher pain intensity.

SECONDARY OUTCOMES:
Summed Pain Intensity Difference Within The First 2 Hours、4 Hours、6 Hours、12 Hours、18 Hours (SPID2、SPID4、SPID6、 SPID12、SPID18) | 0 to 2 hours、0 to 4 hours、0 to 6 hours、0 to 12 hours、0 to 18 hours
  Pain intensity will be evaluated using an 11-point (0-10) numeric rating scale (NRS), with higher numbers indicating a higher pain intensity.
Estimated Time From The Start Of The Infusion Of Study Drug To The First NRS reaching 3 or less | 0 to 24 hours
Total Pain Relief Within The First 2 Hours、4 Hours、6 Hours、12 Hours、18 Hours、24 Hours | 0 to 2 hours、0 to 4 hours、0 to 6 hours、0 to 12 hours、0 to 18 hours、0 to 24 hours
  Patients reported their pain relief using a 5-point(0-4) categorical scale (PR), with "0" indicating "No Relief", "1" indicating "A Little Relief", "2" indicating "Some Relief ", "3" indicating "A Lot of Relief" and "4" indicating "Complete Relief".
Total consumption of remedial analgesics from 0 to 24 hours | 24-hours
Participant' Satisfaction Score For Analgesia Treatment | 24-hours
Investigator Satisfaction Score For Analgesia Treatment | 24-hours
Numbers of Participants With Abnormal Vital Signs | Day 3 or Day 4
  Changes in vital signs such as body temperature (using the celsius system) will be assessed at specified times.
Numbers of Participants With Abnormal Vital Signs | Day 3 or Day 4
  Changes in vital signs such as, blood pressure (using mmHg) will be assessed at specified times.
Numbers of Participants With Abnormal Vital Signs | Day 3 or Day 4
  Changes in vital signs such as , heart rate (measured by beats per minute) will be assessed at specified times.
Numbers of Participants With Abnormal Laboratory Values | Day 3 or Day 4
  Participants with clinically significant lab values will be compared to those receiving placebo comparator.

IPD SHARING:
Plan to Share IPD: Undecided